CLINICAL TRIAL: NCT02199574
Title: Pharmacokinetic Evaluation of EXPAREL in Adults Undergoing Tonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-401
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EXPAREL (Experimental): Single administration of EXPAREL 133 mg (10 mL).
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: EXPAREL — 133 mg EXPAREL in 10 mL.
  Other Names: bupivacaine liposome injectable suspension

SUMMARY:
The purpose of this study is to characterize the pharmacokinetic (PK) profile of a single dose of EXPAREL (133 mg/10 mL) administered intraoperatively per normal infiltration for prolonged analgesia in 12 adult subjects undergoing tonsillectomy with or without removal of the adenoids.

DETAILED DESCRIPTION:
Blood samples for bupivacaine PK analysis will be obtained from subjects at baseline (within 30 minutes prior to EXPAREL infiltration), 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 36, 48, and 72 hours after the beginning of EXPAREL infiltration, and on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years of age at the Screening Visit.
* Subjects undergoing tonsillectomy with or without removal of the adenoids.
* Able and willing to comply with all study visits and procedures.
* Willing and capable of providing written informed consent.

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics.
* Received any investigational drug within 30 days prior to EXPAREL administration, and/or has planned administration of another investigational product or procedure while participating in this study.
* Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after EXPAREL administration. Female subjects must be surgically sterile, at least 2 years postmenopausal, or using an acceptable method of birth control. If of childbearing potential, must have a documented negative pregnancy test within 24 hours before EXPAREL administration.
* Subjects with significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to EXPAREL and/or procedures, or cause inability to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Minkowitz, MD, Principal Investigator — Herman Memorial Hospital, Houston TX
Locations (2):
- United States (2):
  - Memorial Hermann - Memorial City Medical Center, Houston, Texas
  - Memorial Village Surgery Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- EXPAREL: Single administration of EXPAREL 133 mg (10 mL).
  EXPAREL
Period: Overall Study
Arm/Group | EXPAREL
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 11 participants received 133 mg/10 mL EXPAREL following protocol amendment subsequent to 1 participant receiving 266 mg/20 mL EXPAREL according to the original protocol.
Groups:
- EXPAREL: Single administration of EXPAREL 133 mg (10 mL).
  EXPAREL: Protocol was amended after a single subject received a dose of 266 mg EXPAREL to a dose level of 133 mg EXPAREL.
Arm/Group | EXPAREL
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (13.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: From time of study drug administration through Day 7 postdose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EXPAREL
Number analyzed (Participants) | 11
ng/mL | 254 (82.6)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Time Frame: From time of study drug administration through Day 7 postdose
Measure: Median (Full Range); unit: hours
Arm/Group | EXPAREL
Number analyzed (Participants) | 11
hours | 0.50 [0.22 to 35.7]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC(0-t))
Time Frame: From time of study drug administration through Day 7 postdose
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | EXPAREL
Number analyzed (Participants) | 11
hours*ng/mL | 7150 (3189)

4. Primary Outcome: Apparent Terminal Elimination Half-life
Time Frame: From time of study drug administration through Day 7 postdose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | EXPAREL
Number analyzed (Participants) | 3
hours | 9.34 (2.31)

5. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC(0-infinity))
Time Frame: From time of study drug administration through Day 7 postdose
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | EXPAREL
Number analyzed (Participants) | 3
hours*ng/mL | 6379 (2825)

6. Primary Outcome: The Apparent Terminal Elimination Rate Constant (λz)
Time Frame: From time of study drug administration through Day 7 postdose
Measure: Mean (Standard Deviation); unit: 1/hours
Arm/Group | EXPAREL
Number analyzed (Participants) | 3
1/hours | 0.07779 (0.02222)

ADVERSE EVENTS:
Arm/Group | EXPAREL
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXPAREL (N=12)
pyrexia (General disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No